CLINICAL TRIAL: NCT03510208
Title: Phase I/II, Open-Label Study Evaluating the Efficacy and Pharmacokinetics of Panitumumab-IRDye800 as an Optical Imaging Agent to Detect Neoplasms During Neurosurgical Procedures
Brief Title: Panitumumab-IRDye800 in Diagnosing Participants With Malignant Glioma Undergoing Surgery
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-43179; NCI-2018-00536 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRNCNS0009 (Other: Stanford Cancer Institute Palo Alto); R01CA190306 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-04-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Malignant Brain Neoplasm; Malignant Glioma
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (4):
- Cohort 1 -50mg panitumumab-IRDye800 (Experimental): A panitumumab-IRDye800 dose of 50mg (Cohort 1) with or without a 100 mg loading dose of unlabeled panitumumab will be injected 1 to 5 days before the planed standard of care surgery. Participants then undergo NIR imaging during standard of care surgery 1-5 days after receiving panitumumab-IRDye800.
  Interventions: Procedure: Near-Infrared Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800; Device: POINPOINT-IR9000
- Cohort 2 -100mg panitumumab-IRDye800 (Experimental): A panitumumab-IRDye800 dose of 100mg (Cohort 2) with or without a 100 mg loading dose of unlabeled panitumumab will be injected 1 to 5 days before the planed standard of care surgery. Participants then undergo NIR imaging during standard of care surgery 1-5 days after receiving panitumumab-IRDye800.
  Interventions: Procedure: Near-Infrared Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800; Device: POINPOINT-IR9000
- Cohort 3 -100mg panitumumab-IRDye800 (Experimental): Cohort 3 dose will be determined based on Cohort 1 and Cohort 2, with or without a 100 mg loading dose of unlabeled panitumumab will be injected 1 to 5 days before the planed standard of care surgery
  Interventions: Procedure: Near-Infrared Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800; Device: POINPOINT-IR9000
- Cohort 4 (Experimental): Cohort 4 will enroll 24 participants with vestibular schwannomas at the optimal dose of 100mg, as determined by the research team based on data analysis from the first two cohorts.
  Interventions: Procedure: Near-Infrared Fluorescence Imaging; Biological: Panitumumab; Drug: Panitumumab-IRDye800; Device: POINPOINT-IR9000

INTERVENTIONS:
Procedure: Near-Infrared Fluorescence Imaging — Undergo NIR imaging
  Other Names: NIR Fluorescence Imaging; NIR Optical Imaging
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix
Drug: Panitumumab-IRDye800 — Given IV
  Other Names: Panitumumab IRDye 800; RDye800-Panitumumab Conjugate
Device: POINPOINT-IR9000 — Intraoperative camera capable of exciting and detecting near infrared (NIR) dyes. Imaging will be performed on subjects during surgery and/or on ex-vivo resected tissues in the surgery suite ("back table").

SUMMARY:
The phase I/II trial studies the side effects and best dose of panitumumab-IRDye800 in diagnosing participants with malignant glioma who undergo surgery. Panitumumab-IRDye800 can attach to tumor cells and make them more visible using a special camera during surgery, which may help surgeons better distinguish tumor cells from normal brain tissue and identify small tumors that cannot be seen using current imaging methods.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine/verify the safety and pharmacokinetic profile of panitumumab conjugated to the optical dye IRDye800CW (panitumumab-IRDye800), as an imaging agent in patients undergoing surgery for malignant glioma.

SECONDARY OBJECTIVES:

I. Determine the efficacy of panitumumab IRDye800 in identifying malignant glioma compared to surrounding normal central nervous system tissue.

II. Determine whether a loading dose of panitumumab is necessary to achieve an effective tumor-to-background ratio.

III. Determine the optimal timing of the surgical procedure to maximize the tumor-to-background ratio.

OUTLINE: This is a phase I, dose escalation study of panitumumab-IRDye800 followed by a phase II study.

ELIGIBILITY:
Inclusion Criteria:

1) One of the following:

1. Cohorts 1, 2, and 3: Participants with suspected or confirmed diagnosis of glioblastoma
2. Cohort 4: Participants with suspected or confirmed diagnosis of vestibular schwannoma

   2.) Planned surgical removal of the tumor as part of standard of care. This may include participants postchemotherapy, post-radiation, and/or participants who have undergone diagnostic biopsy for their original diagnosis and are felt to be candidates for resection.

   3) Participant age ≥ 18 years.

   4) Participants or their designated advocates must be willing to and capable of providing informed consent and willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

1. Received an investigational drug within 30 days prior to first dose of Panitumumab-IRDye800.
2. Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease as determined by PI; or unstable angina within 6 months prior to enrollment.
3. History of infusion reactions to monoclonal antibody therapies
4. Pregnant or breastfeeding.
5. Evidence of QTc prolongation on pretreatment ECG (greater than 440 ms in males or greater than 460 ms in females).
6. Any of the following lab values:

   1. Platelet count < 75,000/mm3
   2. TSH ≥ 13 micro International Units/mL.
   3. Magnesium, potassium, or calcium < each respective upper limit of normal
   4. Serum creatinine > 1.5 times upper limit of normal
7. Participants receiving Class IA (quinidine, procainamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
8. Participants with a history or evidence of interstitial pneumonitis or pulmonary fibrosis.
9. Participants not deemed by PI to be appropriate candidates for optimal resection of tumor based on location, involvement of eloquent brain, satellite lesions, or other factors not specifically listed here.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of grade 2 or higher adverse events which have been determined to be clinically significant and definitely, probably, or possibly related to the study treatment, graded according to Common Terminology Criteria for Adverse Effects (CTCAE) v. 4.0 | Up to 30 days
  Descriptive statistical analysis of subject disposition, baseline characteristics, exposure to study drug, and adverse events will be performed. Descriptive statistics for continuous data will include mean, standard deviation, median, minimum, maximum, and inter-quartile values. Frequencies and percentages will be used to summarize categorical data.

SECONDARY OUTCOMES:
Tumor to background ratio (TBR) | 30 days from study treatment
  TBR is defined as the fluorescence intensity of tumor tissue compared to that or normal surrounding tissue as determined by ex vivo pathological imaging. Will be analyzed with the individual specimen as the unit of analysis using the Wilcoxon signed rank test.
Panitumumab Loading Dose | 30 days
  The fluorescence intensity of tissue obtained from patients undergoing surgery will be evaluated as an indicator of whether or not the loading dose of panitumumab is necessary to achieve an effective tumor-to-background ratio (TBR). The Fluorescence intensity of tissue will be assessed on the specimens collected on the day of surgery (Day 1-5 Post infusion), in group a vs group b, for Cohorts 1 and 2, in order to determine the tumor-to-background ratio (TBR). The outcome will be expressed as TBR by group and cohort. TBR will be reported as means +/- STD.
Optimal Timing of Surgical Procedure | 1 year
  The fluorescence intensity of tissue collected at surgery will be measured 1 to 5 days after infusion, and the outcome will be assessed as highest daily mean tumor-to-background ratio (TBR), with standard deviation. The tissue analysis to obtain the outcome data will occur within 1 year from surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Li, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No